CLINICAL TRIAL: NCT05388097
Title: A Novel Strategy for Addressing Social Barriers to a Successful, Sustained Discharge From the Hospital for Acute Heart Failure
Brief Title: Effect of a Quality Improvement Initiative to Address Social Determinants of Health on Rehospitalization Rates in Patients With Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Collaborators: Truman Medical Center (Other); University of Missouri, Kansas City (Other); Mid America Regional Council (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Managed Services Network
Record Dates: First submitted 2022-04-27; First posted 2022-05-24 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure
Keywords: heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Of Care - No Managed Services (No Intervention): Subjects receive standard medical care and follow-up after hospital discharge
- Managed Services After Discharge (Experimental): Subjects receive in-home assessment and care coordination/connection with community resources after hospital discharge
  Interventions: Other: Managed Services

INTERVENTIONS:
Other: Managed Services — coordination of care and assistance with community resources (food, transportation)
  Arms: Managed Services After Discharge

SUMMARY:
The objective of this program is to improve post-acute care coordination for necessary social services for patients leaving the hospital after recovering from an episode of decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-99 years
* Resident of Missouri or Kansas
* Current inpatient admission for acute heart failure

Exclusion Criteria:

* Under 18 years or over 99 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in all-cause re-hospitalization | 2 years
  reduction in all-cause re-hospitalization via improved post-acute care coordination

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Olathe Health System, Olathe, Kansas
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Curators of the University of Missouri. University of Missouri-Kansas City Community Connect: Doing More Together. — https://community.umkc.edu/about/
- See also: University of Missouri-Kansas City (UMKC). School of Education. — https://education.umkc.edu/outreach-research/
- See also: Truman Medical Centers-Health Sciences District. Community Health Needs Assessment. June 2019. — https://res.cloudinary.com/dpmykpsih/image/upload/truman-site-261/media/7535ea7dec474654bdf95f9e7ef463cb/tmc-hospital-hill-2019-final-2.pdf
- See also: Truman Medical Center Foundation — https://www.tmcgiving.org/our-mission/